CLINICAL TRIAL: NCT01404169
Title: A 24-weeks, Multi-center, Randomized, Double-blind, Placebo Controlled Study to Evaluate the Efficacy and Safety of Donepezil Hydrochloride in Chinese Subjects With Severe Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E2020-C086-339
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Type Dementia
Keywords: Alzheimer Disease; Dementia; Delirium; Amnestic; Cognitive Disorders; Donepezil; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders; Cholinesterase Inhibitors; Enzy
MeSH Terms: conditions — Alzheimer Disease; Dementia; Delirium; Cognitive Dysfunction; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: E2020
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2020 — In titration period, donepezil 5-mg tablet will be taken orally once daily for 6 weeks, following donepezil 10 mg tablets taken orally once daily for 18 weeks in the maintenance period.
  Arms: 1
Drug: Placebo — Placebo matched to donepezil 5 mg or 10 mg tablets taken orally once daily for 24 weeks.
  Arms: 2

SUMMARY:
The objective is to demonstrate that donepezil hydrochloride 10 mg/day has superior efficacy compared with placebo in cognitive function in Chinese subjects with severe Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria

* Written informed consent (IC) will be obtained from the subject (if possible) or from the subject's legal guardian or legal representative prior to beginning screening activities.
* Subject age range: male and female subjects 50 to 90 years of age, inclusive
* Diagnosis: diagnostic evidence of probable Alzheimer's Disease (AD) consistent with Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) and National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* MMSE 1 to 12 inclusive, at both Screening and Baseline
* SIB less than or equal to 90 and greater than or equal to 10 at both Screening and Baseline
* Comorbid medical conditions must be clinically stable prior to Baseline, unless otherwise specified.

Exclusion Criteria

* Subjects with a known history of disorders that affect cognition or the ability to assess cognition, but are distinguishable from AD
* Evidence of focal disease to account for dementia on any cranial image MRI or CT.
* Subjects with dementia complicated by other organic disease or AD with delirium according to DSM-IV criteria
* Subjects who cannot swallow or who have difficulty swallowing whole tablets, as tablets should not be broken or crushed
* Illiteracy prior to AD
* Subjects who are unwilling or unable to fulfill the requirements of the study
* Treatment with another cholinesterase inhibitor and/or memantine in the 3 months prior to Screening
* Subjects with a poor response (tolerability) to prior exposure to donepezil

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The change in the total Severe Impairment Battery (SIB) score at Week 24 | 24 weeks
  All statistical tests will be conducted at the 0.05 level of significance (two-tailed). A positive outcome will be declared if for the primary efficacy endpoint as measured by the Severe Impairment Battery (SIB), the change from Baseline to Week 24 in the total SIB score last observation carried forward (LOCF) demonstrates superiority for donepezil 10 mg, compared with placebo.

SECONDARY OUTCOMES:
Clinician Interview-Based Impression of Severity (CIBIC)+ overall score at Week 24 | 24 weeks
  An ANCOVA with embedded Cochran-Mantel-Haenszel (CMH) test will be used with the CIBIC+ and center in the model. Overall change from Baseline in scores at Week 24 (LOCF) will be analyzed with the same model as the SIB.

CONTACTS AND LOCATIONS:
Overall Officials: Naoki Kubota, Study Director — Neuroscience Clinical Development Section, Japan/Asia Clinical Research Product Creation Unit, Eisai Co., Ltd.
Locations (32):
- China (32):
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Huilongguan Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangzhou Brain Hospital, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Union Hospital, Tongji Medical college Huazhong University of Science and Technology, Wuhan, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of YueYang, Yueyang, Hunan
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong
  - Hushan Hospital affliated to Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, The Fourth Military Medical University, Xi’an, Shanxi
  - Xi'An Mental Health Center, Xi’an, Shanxi
  - Xijing Hospital, The Fourth Military Medical University, Xi’an, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Nanjing Brain Hospital, Nanjing Jiangsu
  - Tianjin Anding Hospital, Tianjin
  - Tianjin People's Hospital, Tianjin